CLINICAL TRIAL: NCT00583739
Title: Effect of a Yoga Intervention on Fatigue, Distress, and Quality of Life in Breast Cancer Patients: A Randomized Pilot Study
Brief Title: Yoga to Reduce Cancer Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Geraldine Jacobson, MD, MPH, Department of Radiation Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 200707733
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Breast Neoplasm
Keywords: Fatigue; Yoga; Anxiety; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Yoga intervention
  Interventions: Behavioral: Yoga
- 2 (No Intervention): Control. No Yoga for 8 weeks.

INTERVENTIONS:
Behavioral: Yoga — Gentle Yoga for breast cancer survivors, 1 time weekly, for 8 weeks.
  Arms: 1

SUMMARY:
A randomized trial from the British National Health Service found that supervised exercise benefits women with early stage breast cancer with improved functional and psychological benefit after a 12-week intervention and 6 months later. Considering the needs of breast cancer patients and survivors and the reported benefits of exercise and yoga intervention, the investigators propose a pilot study of an 8-week yoga intervention in breast cancer patients. This study would specifically address measures of fatigue and psychosocial distress in the population of breast cancer patients during treatment and within the year following treatment. Currently there is very limited literature on yoga intervention in this population.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must have had histologically or cytologically confirmed breast cancer. This includes, but is not limited to: breast cancer-in situ; ductal carcinoma in situ; lobular carcinoma in situ; cystosarcoma phyllodes; inflammatory breast carcinoma; invasive breast carcinoma; and breast cancer not otherwise specified; cancer must be stage 0 through stage III.
* Treatment completion within the past calendar year.
* Age ≥ 18 years. While breast cancer can occur in the pediatric population, the pediatric population is best served by trials specifically designed for their age group.
* Life expectancy of greater than 1 year.
* Karnofsky ≥ 60%; see Appendix A.
* Women of childbearing potential are eligible for this study.
* Pregnant women are eligible for this study pending a doctor's note.
* The ability to understand and complete the study questionnaires.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with known metastasis.
* Patients who are actively participating in a yoga class.
* Known uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would compromise subject health during yoga.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Determine if an 8 week yoga program designed for breast cancer patients improves subjective reports of overall well being and fatigue | 8 weeks

SECONDARY OUTCOMES:
Analyze symptoms of depression and anxiety | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Jacobson, MD MPH, Principal Investigator — department of radiation oncology
Locations (1):
- The University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Bower JE, Woolery A, Sternlieb B, Garet D. Yoga for cancer patients and survivors. Cancer Control. 2005 Jul;12(3):165-71. doi: 10.1177/107327480501200304. PMID 16062164
- [Background] Culos-Reed SN, Carlson LE, Daroux LM, Hately-Aldous S. A pilot study of yoga for breast cancer survivors: physical and psychological benefits. Psychooncology. 2006 Oct;15(10):891-7. doi: 10.1002/pon.1021. PMID 16374892